CLINICAL TRIAL: NCT04510649
Title: Ph. 1, Open-label, 2 Part, 2 Period Fixed-Sequence Crossover Study to Assess the Effect of Rabeprazole, a Proton Pump Inhibitor, and the Effect of Rifampin, a Strong CYP3A Inducer, on the Pharmacokinetics of Surufatinib in Healthy Subjects
Brief Title: Surufatinib DDI With a PPI and a CYP3A Inducer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hutchison Medipharma Limited (Industry)
Responsible Party: Sponsor
Organization: Hutchmed (Industry)
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 2020-012-00US1
Record Dates: First submitted 2020-08-10; First posted 2020-08-12 (Actual); Last update posted 2021-06-18 (Actual); Status verified 2020-08

CONDITIONS: Healthy
MeSH Terms: interventions — Rabeprazole; Medicare Part B; Rifampin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Surufatinib and Rabeprazole (Part A) (Experimental): Part A: Surufatinib 300 mg on study days 1 and 11 Rabeprazole 40 mg on study days 5 - 11
  Interventions: Drug: Part A
- Surufatinib and Rifampin (Part B) (Experimental): Part B: Surufatinib 300 mg on study days 1 and 12 Rifampin 600 mg on study days 5-15
  Interventions: Drug: Part B

INTERVENTIONS:
Drug: Part A — in Part A, all subjects will receive Surufatinib 300 mg in a single dose on study days 1 and 11 and receive Rabeprazole 30 mg single dose on study days 5 through 11
  Other Names: Rabeprazole 30 mg
  Arms: Surufatinib and Rabeprazole (Part A)
Drug: Part B — in Part B, all subjects will receive Surufatinib 300 mg in a single dose on study days 1 and 12 and receive Rifampin 600 mg single dose on study days 5 through 16
  Other Names: Rifampin 600 mg
  Arms: Surufatinib and Rifampin (Part B)

SUMMARY:
The purpose of this is to evaluate the effect of proton pump inhibitor (rabeprazole) and the effect of a CYP3A inducer (rifampin) on the pharmacokinetics of Surufatinib.

DETAILED DESCRIPTION:
This study will be a single center, open-label, 2 part, 2 period fixed-sequence crossover study to be conducted with 28 healthy male and female subjects (part A and part B). Subjects will be enrolled in either part A or part B.

In Part A, subjects will be administered surufatinib alone in treatment Period 1 and co-administered with rabeprazole in treatment Period 2.

In Part B, subjects will be administered surufatinib alone in treatment Period 1 and co-administered with rifampin in treatment Period 2.

PK samples will be collected through out both study periods.Subjects will be confined in the clinic from check-in on Day -1 through the end-of study visit on Day 15 (part A) and Day 16 (part B).

ELIGIBILITY:
Inclusion Criteria

* Non-smoking, healthy male or female between the ages of 18 and 55 years (inclusive)
* Body mass index (BMI) > 18 and ≤ 29 kg/m2
* Females must be of non-childbearing potential or surgically sterile
* Males who have not had a successful vasectomy and are partners of women of childbearing potential must use, or their partners must use, a medically acceptable method of contraception starting for at least 1 menstrual cycle prior to and throughout the entire study period, and for 2 weeks after the last dose of study drug. Those with partners using hormonal contraceptives must also use an additional approved method of contraception such as a condom with spermicide. Males who have had a successful vasectomy (confirmed azoospermia, documentation needed) require no additional contraception. No sperm donation is allowed during the study period and for 90 days after study drug discontinuation.

Exclusion Criteria

* Evidence of clinically significant cardiovascular, hepatic, GI, renal, respiratory, endocrine, hematological, neurological, or psychiatric disease or abnormalities
* Known history of any GI surgery or any condition possibly affecting drug absorption, however appendectomy and hernia repair will be allowed
* Clinically significant illness within 8 weeks or a clinically significant infection within 4 weeks prior to first dose
* Known food allergy deemed clinically significant.
* Clinically significant deviation from normal in the physical examination, vital signs, or clinical laboratory determinations
* Systolic blood pressure > 140 mmHg or diastolic blood pressure > 90 mmHg
* Clinically significant ECG abnormality, including a marked baseline prolongation of QT/QTc interval (eg, repeated demonstration of a QTcF interval > 480 msec), or had a family history of prolonged QTc syndrome or sudden death
* Has Gilbert's syndrome as indicated by total bilirubin > upper limit of normal (ULN) and subsequent measurement of direct bilirubin is not within normal range.
* History of smoking or use of nicotine-containing substances within the previous 2 months
* History of drug or alcohol misuse in the previous 6 months
* Diagnosed with acquired immune deficiency syndrome (AIDS) or has performed tests that are positive for human immunodeficiency virus (HIV), Hepatitis B virus (HBV), or Hepatitis C virus (HCV)
* Participated in a clinical trial of other drug and the last use of other study drug is less than 5 times the half-life or 4 weeks, whichever is longer, or the subject is currently enrolled in another clinical trial
* Consumes grapefruit, starfruit, Seville oranges, or their products within 7 days before first dose
* Consumes herbal preparations/medications, including, but not limited to kava, ephedra (ma huang), Ginkgo biloba, dehydroepiandrosterone (DHEA), yohimbe, saw palmetto, and ginseng within 7 days before first dose
* Weight loss or gain of > 10% within 4 weeks before first dose
* Received blood or blood products within 4 weeks, or donated blood or blood products within 8 weeks, or donated double red blood cells within 16 weeks before first dose
* Uses any over-the-counter (OTC) medications or prescription drugs within 2 weeks before first dose
* Uses CYP3A inducers (including St. John's wort) or inhibitors within 2 weeks before first dose
* Allergic to the study drugs (including rabeprazole or rifampin) or to any of the excipients
* Cannot abstain from using a proton pump inhibitor (PPI) or a histamine H2 receptor antagonist (H2 blocker) or locally acting antacids (eg, Gaviscon, Gelusil, Maalox, Milk of Magnesia, Mylanta, Rolaids, Tums)
* Female participant is pregnant, lactating, or breastfeeding

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2020-07-09 (Actual); Primary Completion 2020-09-11 (Actual); Study Completion 2021-03-02 (Actual)

PRIMARY OUTCOMES:
AUC (0-t) of Surufatinib [ Time Frame: Up to Day 15 ] Pharmacokinetics of surufatinib by assessment of area under the plasma concentration time curve from zero to the last measurable concentration | up to 16 days
  Pharmacokinetics of surufatinib by assessment of area under the plasma concentration time curve from zero to the last measurable concentration
AUC of Surufatinib | up to 16 days
  Pharmacokinetics of surufatinib by assessment of area under the plasma concentration curve from zero extrapolated to infinity (if data permit)
Cmax of Surufatinib | up to 16 days
  Pharmacokinetics of Surufatinib by assessment of maximum plasma Surufatinib concentration

SECONDARY OUTCOMES:
Number of participants with treatment emergent adverse events as assessed by CTCAE v5.0 | up to 16 days
  To evaluate the safety, in healthy subjects, of a single dose of 300 mg surufatinib administered alone and with rabeprazole or rifampin

CONTACTS AND LOCATIONS:
Overall Officials: Youngiun Kim, MD, Principal Investigator — WCCT Global Inc.
Locations (1):
- West Coast Clinical Trials (WCCT), Cypress, California, United States